CLINICAL TRIAL: NCT01874665
Title: Phase 2 Trial of Ponatinib in Patients With Metastatic and/or Unresectable Gastrointestinal Stromal Tumor Following Failure of Prior Tyrosine Kinase Inhibitor Therapy
Brief Title: A Phase 2 Trial of Ponatinib in Participants With Metastatic and/or Unresectable Gastrointestinal Stromal Tumor
Acronym: GIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP24534-12-202
Record Dates: First submitted 2013-05-29; First posted 2013-06-11 (Estimated); Results first posted 2016-05-17 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: GIST
Keywords: Gastrointestinal Neoplasms; Gastrointestinal stromal tumor; mesenchymal tumor
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Stromal Tumors | interventions — ponatinib

ARMS (2):
- Cohort A (Experimental): Participants with KIT exon 11-mutant GIST.
  Interventions: Drug: Ponatinib
- Cohort B (Experimental): Participants with GIST that lack KIT exon 11 mutations (Cohort B).
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib 45 mg, tablets, orally, once-daily.
  Other Names: AP24534; Iclusig

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ponatinib in participants with metastatic and/or unresectable gastrointestinal stromal tumor (GIST) following failure of prior tyrosine kinase inhibitor (TKI) therapy.

DETAILED DESCRIPTION:
This is a non-randomized, open label, multi-center phase 2 study to evaluate the efficacy and safety of ponatinib in participants with metastatic and/or unresectable GIST after failure of prior TKI therapy. Participants whose tumors have an activating mutation in exon 11 of cellular KIT (KIT) will be enrolled into Cohort A. Participants whose tumors have other activating mutations will be enrolled into in Cohort B.

The primary objective is to assess clinical benefit in participants with KIT exon 11-mutant GIST (Cohort A) defined as clinical benefit rate (CBR), which is the composite of complete response (CR), partial response (PR) and stable disease (SD) lasting greater than or equal to (>=) 16 weeks per modified response evaluation criteria in solid tumors (RECIST 1.1) as a measure of disease control. The secondary objective is to assess clinical benefit in participants with GIST that lacks an activating KIT exon 11 mutation (Cohort B) and in the total participant population. The efficacy assessments are tumor response using RECIST Version 1.1, modified for GIST and assessment of progression-free survival (PFS) and overall survival (OS). The safety assessments include routine physical and laboratory evaluations, electrocardiograms (ECGs), echocardiograms (ECHOs), and adverse event (AE) monitoring. Other assessments include optional 18F fluorodeoxyglucose positron emission tomography (FDG-PET); optional pre- and post-treatment tumor biopsy for pharmacodynamic studies; and pharmacokinetics (PK). It is estimated that accrual will be complete within 1 year; the total estimated duration of the study is 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants >=18 years old.
2. GIST with failure of prior TKI therapy defined as:

   1. Histologically confirmed metastatic and/or unresectable GIST after experiencing failure of prior treatment with imatinib, sunitinib, and regorafenib. If prior TKI treatment was neoadjuvant therapy, then relapse must have occurred during the neoadjuvant therapy in order to consider it failed therapy.
   2. Participants in Cohort A must have evidence of activation mutations in exon 11 of KIT in their tumors. Demonstration of an exon 11 mutation may be based on prior assessment or on evaluation of a tumor sample after enrollment in this study. Participants in Cohort B must have GIST that lacks activating mutations in KIT exon 11, but may have evidence of another activating mutation such as in KIT exon 9 or in PDGFR-α. Participants may be enrolled in the study prior to determination of the appropriate cohort (as long as both cohorts are open for enrollment).
3. Measurable disease per modified RECIST 1.1. A lesion in a previously irradiated area is eligible to be considered as measurable disease as long as there is objective evidence of progression of the lesion prior to study enrollment.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
5. Adequate hepatic function as defined by the following criteria:

   1. Total serum bilirubin less than or equal to (<=) 1.5*Upper Limit of Normal (ULN), unless due to Gilbert's syndrome.
   2. ALT <=2.5*ULN or <=5.0*ULN if liver metastases are present.
   3. AST <=2.5*ULN or <=5.0*ULN if liver metastases are present.
6. Adequate renal function as defined by the following criterion:

   a. Serum creatinine <1.5*ULN.
7. Adequate pancreatic function as defined by the following criterion:

   a. Serum lipase and amylase <=1.5*ULN.
8. For participants of childbearing potential, a negative pregnancy test must be documented prior to enrollment.
9. Female and male participants who are fertile must agree to use an effective form of contraception with their sexual partners from signing of the informed consent form for this study through 4 months after the end of treatment.
10. Provision of written informed consent.
11. Willingness and ability to comply with scheduled visits and study procedures
12. Fully recovered (<= Grade 1 or returned to baseline or deemed irreversible) from the acute effects of prior cancer therapy before initiation of study drug.

Exclusion Criteria:

1. Major surgery within 28 days prior to initiating therapy
2. History of bleeding disorder
3. History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
4. History of alcohol abuse
5. Uncontrolled hypertriglyceridemia (triglycerides >450 milligram per deciliter [mg/dL])
6. Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   1. Any history of myocardial infarction (MI).
   2. Any history of unstable angina.
   3. Congestive heart failure within 6 months prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards within 6 months prior to enrollment.
   4. History of clinically significant (as determined by the treating physician) atrial arrhythmia.
   5. Any history of ventricular arrhythmia.
   6. Any history of cerebrovascular accident or transient ischemic attack (TIA).
   7. Any history of peripheral vascular infarction, including visceral infarction; or any revascularization procedure of any vasculature, including the placement of a stent.
   8. Venous thromboembolism including deep venous thrombosis (DVT) or pulmonary embolism within 6 months prior to enrollment.
7. Uncontrolled hypertension (diastolic blood pressure greater than (>) 90 millimeter of mercury [mmHg]; systolic >150 mmHg). Participants with hypertension should be under treatment on study entry to effect blood pressure control.
8. Taking medications with a known risk of Torsades de Pointes.
9. Taking any medications or herbal supplements that are known to be strong inhibitors of cytochrome P3A4 (CYP3A4) within at least 14 days before the first dose of ponatinib.
10. Ongoing or active infection. This includes but is not limited to the requirement for intravenous antibiotics.
11. Known history of human immunodeficiency virus (HIV). Testing is not required in the absence of prior documentation or known history.
12. Pregnant or breastfeeding.
13. Malabsorption syndrome or other gastrointestinal illness that could affect oral absorption of study drugs.
14. Individuals with a history of a different malignancy, other than cervical cancer in situ, basal cell or squamous cell carcinoma of the skin, are ineligible, except if they have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy OR if the other primary malignancy is neither currently clinically significant nor requiring active intervention.
15. Use of any approved TKIs or investigational agents within 2 weeks or 6 half-lives of the agent, whichever is longer, prior to receiving study drug.
16. Any condition or illness that, in the opinion of the investigator, would compromise participant safety or interfere with the evaluation of the drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-06-05 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2016-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Site #047, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Site #008, Boston, Massachusetts
  - Oregon Health & Sciences University, Site #048, Portland, Oregon
  - Fox Chase Cancer Center, Site #012, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Participants with KIT exon 11-mutant GIST ponatinib: 45 milligram (mg), taken orally once-daily.
- Cohort B: Participants with gastrointestinal stromal tumors (GIST) that lack KIT exon 11 mutations (Cohort B) ponatinib: 45 mg, taken orally once-daily.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 30 | 15
Completed | 0 | 0
Not Completed | 30 | 15
Not completed — Adverse Event | 6 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Clinical Progressive Disease | 4 | 3
Not completed — Study Terminated by Sponsor | 0 | 2
Not completed — Documented Progressive Disease | 11 | 7
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: The intention to treat (ITT) population included all participants who received any dose of ponatinib in the study.
Groups:
- Cohort A: Participants with KIT exon 11-mutant GIST ponatinib: 45 mg, taken orally once-daily.
- Cohort B: Participants with GIST that lack KIT exon 11 mutations (Cohort B) ponatinib: 45 mg, taken orally once-daily.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The ITT population included all participants who received any dose of ponatinib in the study.
  years | 59.3 (10.37) | 53.9 (16.06) | 57.5 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The ITT population included all participants who received any dose of ponatinib in the study.
  Participants
    Female | 11 | 8 | 19
    Male | 19 | 7 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT population included all participants who received any dose of ponatinib in the study.
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 29 | 15 | 44
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT population included all participants who received any dose of ponatinib in the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 29 | 15 | 44
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: The ITT population included all participants who received any dose of ponatinib in the study.
  Participants
    United States | 30 | 15 | 45
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The ITT population included all participants who received any dose of ponatinib in the study.
  kilogram (kg) | 80.12 (20.699) | 75.10 (13.917) | 78.45 (18.702)
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The ITT population included all participants who received any dose of ponatinib in the study.
  centimeter (cm) | 171.20 (7.839) | 171.28 (7.149) | 171.23 (7.534)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) in Cohort A
Description: To assess clinical benefit rate in participants with KIT exon 11-mutant GIST.It is defined as the composite of complete response(CR),partial response(PR),and stable disease(SD) lasting >=16 weeks per modified Response Evaluation Criteria In Solid Tumors(RECIST) 1.1 as a measure of disease control.CR is complete disappearance of all target lesions and non-target disease, with the exception of nodal disease.All nodes, both target and non-target, must decrease to normal (short axis <10millimeter [mm]).No new lesions.PR is >=30% decrease under baseline of the sum of diameters of all target lesions.The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions.No unequivocal progression of non-target disease.No new lesions.SD is not qualifying for CR,PR,Progressive Disease(PD).PD is >=20% increase from the smallest prior sum of the longest diameter(SLD)and with >=5mm absolute increase, or appearance of a new lesion.
Time Frame: 16 weeks after first dose
Population: The ITT population included all participants who received any dose of ponatinib in the study. The ITT population where data at specified time points was available.
Measure: Number (95% Confidence Interval); unit: percentage (%) of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 28
percentage (%) of participants | 35.7 [18.6 to 55.9]

2. Secondary Outcome: Clinical Benefit Rate (CBR) in Cohort B
Description: To assess clinical benefit rate in participants with GIST that lacks KIT exon 11 mutations (Cohort B) and in the total participant population. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 millimeter [mm]). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. SD was defined as not qualifying for CR, PR, PD.
Time Frame: 16 weeks after first dose
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Number (95% Confidence Interval); unit: percentage (%) of participants
Arm/Group | Cohort B
Number analyzed (Participants) | 15
percentage (%) of participants | 20.0 [4.3 to 48.1]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of study drug administration to time of objective disease progression or death due to any cause, whichever may come first. To assess PFS in each cohort and in the total participant population.
Time Frame: From date of enrollment until the end of the study or disease progression or death due to any cause, whichever came first, assessed up to 3 years
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 30 | 15
days | 112.0 [57.0 to 252.0] | 57.0 [55.0 to 502.0]

4. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: ORR is defined as the composite of CR and PR per Response Evaluation Criteria in RECIST 1.1, assessed for each cohort and in the total participant population. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions.
Time Frame: From date of enrollment until discontinuation or the end of the study, whichever came first, assessed up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 28 | 15
percentage of participants | 7.1 [0.9 to 23.5] | 0.0 [0.0 to 21.8]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time interval between the first dose of study drug to death due to any cause. Overall survival was analyzed using the Kaplan-Meier method.
Time Frame: From first dose of drug until the end of the study or death, whichever came first, assessed up to 3 years
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 30 | 15
days | 411.0 [234.0 to 836.0] | 399.0 [90.0 to NA] — Upper limit of confidence interval was not estimable.

6. Secondary Outcome: Number of Participants With Physical Examination
Time Frame: From date of enrollment until the End-of-Treatment, assessed up to 3 years
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 30 | 15
Participants | 6 | 1

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Vital Sign Measurements
Time Frame: From date of enrollment until the End-of-Treatment, assessed up to 3 years
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 30 | 15
Participants
  Hypertension | 15 | 2
  Procedural hypotension | 1 | 0
  Pyrexia | 7 | 3
  Chills | 3 | 1
  Feeling of body temperature change | 1 | 0

8. Secondary Outcome: Number of Participants With Worst Shift From Baseline Values to Post-baseline Values in Laboratory Parameters
Time Frame: From date of enrollment until the End-of-Treatment, assessed up to 3 years
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 30 | 15
Participants
  Albumin decreased | 13 | 4
  Alkaline phosphatase increased | 12 | 8
  Alanine aminotransferase (ALT) increased | 11 | 7
  Amylase | 3 | 5
  Absolute neutrophil count (ANC) decreased | 2 | 0
  Aspartate aminotransferase (AST) increased | 11 | 8
  Bicarbonate decreased | 1 | 1
  Bilirubin | 4 | 2
  Calcium decreased | 5 | 4
  Calcium increased | 5 | 1
  Creatinine increased | 3 | 3
  Glucose decreased | 1 | 3
  Glucose increased | 19 | 9
  Hemoglobin decreased | 10 | 5
  Lipase increased | 6 | 7
  Lymphocytes (ALC)/ lymphopenia | 5 | 4
  Phosphorus decreased | 5 | 1
  Platelets decreased | 2 | 0
  Potassium decreased | 5 | 2
  Potassium increased | 8 | 3
  Sodium decreased | 8 | 1
  Sodium increased | 7 | 2
  Triglycerides increased | 2 | 0
  White blood cells (WBC) decreased | 2 | 0

9. Secondary Outcome: Number of Participants With TEAEs Related to Electrocardiogram (ECG) Findings
Time Frame: From date of enrollment until the End-of-Treatment, assessed up to 3 years
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 30 | 15
Participants
  Ejection Fraction Decreased | 1 | 2
  Atrial Fibrillation | 1 | 2
  Sinus Tachycardia | 1 | 1
  Cardiac Failure Congestive | 1 | 0
  Myocardial Ischaemia | 1 | 0
  Pericardial Effusion | 0 | 1
  Right Ventricular Dysfunction | 1 | 0
  Sinus Bradycardia | 1 | 0

10. Secondary Outcome: Number of Participants With TEAEs Related to Echocardiography Parameter
Time Frame: From date of enrollment until the End-of-Treatment, assessed up to 3 years
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 30 | 15
Participants
  Congestive Cardiac Failure | 1 | 0
  Right Ventricular Dysfunction | 1 | 0
  Decreased Ejection Fraction | 1 | 2
  Pulmonary Oedema | 0 | 1

11. Secondary Outcome: Number of Participants Reporting One or More TEAEs and Serious Adverse Event (SAE)
Time Frame: From date of enrollment until the End-of-Treatment, assessed up to 3 years
Population: The ITT population included all participants who received any dose of ponatinib in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 30 | 15
Participants
  TEAE | 30 | 15
  SAE | 20 | 6

12. Secondary Outcome: Cmax, SS: Maximum Observed Plasma Concentration at Steady State for Ponatinib
Time Frame: Pre-dose and at multiple timepoints (up to 1 month) post-dose
Population: Data was not collected for Cmax,ss, since outcome measure was not planned to be analyzed.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (up to 3 years)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 4/30 | 2/15
Serious Adverse Events (participants affected / at risk) | 20/30 | 6/15
Other Adverse Events (participants affected / at risk) | 30/30 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=30) | Cohort B (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 1
DUODENAL STENOSIS (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0
SMALL INTESTINAL ULCER PERFORATION (Gastrointestinal disorders) | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 0
FATIGUE (General disorders) | 1 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
COLONIC ABSCESS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 0
SEPSIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=30) | Cohort B (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 5
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 2
HYPOTHYROIDISM (Endocrine disorders) | 3 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 14 | 6
ASCITES (Gastrointestinal disorders) | 3 | 1
CONSTIPATION (Gastrointestinal disorders) | 14 | 5
DIARRHOEA (Gastrointestinal disorders) | 8 | 2
DRY MOUTH (Gastrointestinal disorders) | 3 | 1
DYSPEPSIA (Gastrointestinal disorders) | 4 | 4
NAUSEA (Gastrointestinal disorders) | 6 | 3
STOMATITIS (Gastrointestinal disorders) | 1 | 2
VOMITING (Gastrointestinal disorders) | 7 | 2
CHILLS (General disorders) | 3 | 1
FATIGUE (General disorders) | 15 | 9
NON-CARDIAC CHEST PAIN (General disorders) | 3 | 1
OEDEMA PERIPHERAL (General disorders) | 13 | 3
PAIN (General disorders) | 2 | 1
PYREXIA (General disorders) | 7 | 3
PNEUMONIA (Infections and infestations) | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 1 | 3
FALL (Injury, poisoning and procedural complications) | 2 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 5
AMYLASE INCREASED (Investigations) | 1 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 | 5
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 7 | 6
EJECTION FRACTION DECREASED (Investigations) | 1 | 2
LIPASE INCREASED (Investigations) | 3 | 4
WEIGHT DECREASED (Investigations) | 6 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 11 | 4
DEHYDRATION (Metabolism and nutrition disorders) | 5 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 3
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 15 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
DIZZINESS (Nervous system disorders) | 3 | 2
HEADACHE (Nervous system disorders) | 13 | 7
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 4 | 0
INSOMNIA (Psychiatric disorders) | 4 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 2
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 3 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 | 4
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 3 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 11 | 4
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 3
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 3
RASH (Skin and subcutaneous tissue disorders) | 15 | 12
HYPERTENSION (Vascular disorders) | 15 | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 1 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 0
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
ERUCTATION (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 | 0
PROCTALGIA (Gastrointestinal disorders) | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 0
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1
ORAL INFECTION (Infections and infestations) | 1 | 0
OTITIS MEDIA (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 1
PYURIA (Infections and infestations) | 0 | 1
SKIN INFECTION (Infections and infestations) | 0 | 1
TOOTH INFECTION (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
INCISION SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 | 0
NUCHAL RIGIDITY (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 2
MEMORY IMPAIRMENT (Nervous system disorders) | 2 | 0
TREMOR (Nervous system disorders) | 0 | 2
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
DIZZINESS POSTURAL (Nervous system disorders) | 1 | 0
DYSAESTHESIA (Nervous system disorders) | 1 | 0
HYPERAESTHESIA (Nervous system disorders) | 1 | 0
LETHARGY (Nervous system disorders) | 1 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 2
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | 0
DYSURIA (Renal and urinary disorders) | 0 | 2
MICTURITION URGENCY (Renal and urinary disorders) | 1 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1
NOCTURIA (Renal and urinary disorders) | 1 | 0
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 | 0
URINARY TRACT PAIN (Renal and urinary disorders) | 0 | 1
GYNAECOMASTIA (Reproductive system and breast disorders) | 1 | 0
TESTICULAR PAIN (Reproductive system and breast disorders) | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 2 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0
PITYRIASIS RUBRA PILARIS (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0
RASH FOLLICULAR (Skin and subcutaneous tissue disorders) | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 | 0
FLUSHING (Vascular disorders) | 1 | 1
HOT FLUSH (Vascular disorders) | 1 | 0
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 1 | 2
DIPLOPIA (Eye disorders) | 1 | 0
DRY EYE (Eye disorders) | 1 | 0
EPISCLERITIS (Eye disorders) | 0 | 1
EYELID PAIN (Eye disorders) | 1 | 0
HYPERMETROPIA (Eye disorders) | 1 | 0
PERIORBITAL OEDEMA (Eye disorders) | 1 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 1 | 2
VISUAL IMPAIRMENT (Eye disorders) | 1 | 0
VITREOUS DETACHMENT (Eye disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
EAR DISCOMFORT (Ear and labyrinth disorders) | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 1 | 0
HYPOACUSIS (Ear and labyrinth disorders) | 1 | 0
EARLY SATIETY (General disorders) | 2 | 1
ASTHENIA (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 0
FACE OEDEMA (General disorders) | 1 | 0
FEELING OF BODY TEMPERATURE CHANGE (General disorders) | 1 | 0
MALAISE (General disorders) | 1 | 0
PERIPHERAL SWELLING (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study is ongoing. Uncontrolled Study. Small participant population. Non-randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for up to 1 year (to first generate a multicenter publication) and a period that is 60 to 120 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication to delete confidential information, excluding the results of the Study.